CLINICAL TRIAL: NCT02434055
Title: Evaluation of a Novel Method of Contrast Volume Quantification - The AVERT PLUS
Brief Title: Evaluation of a Novel Method of Contrast Volume Quantification - AVERT PLUS
Acronym: AVERT-PLUS
Status: Terminated | Type: Observational
Why Stopped: Business purposes
Sponsor: Anand Prasad (Other)
Collaborators: Osprey Medical, Inc (Industry)
Responsible Party: Sponsor-Investigator, Anand Prasad, Assistant Professor of Medicine, The University of Texas Health Science Center at San Antonio
Organization: The University of Texas Health Science Center at San Antonio (Other)
Other Study IDs: HSC20150190H
Record Dates: First submitted 2015-04-29; First posted 2015-05-05 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Extravasation of Contrast Media
MeSH Terms: conditions — Extravasation of Diagnostic and Therapeutic Materials

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: AVERT PLUS

SUMMARY:
Purpose: To evaluate the accuracy of the AVERT PLUS to monitor contrast volume used during angiographic procedures.

Research Design: The AVERT PLUS is an FDA 510K cleared device which consists of a contrast delivery modulator designed to reduce unnecessary contrast dye delivery to the patient during angiography (coronary or peripheral) and a concomitant system to precisely measure contrast volume delivered to the patient. This will be a first in man prospective observational study of the accuracy of this system to quantify contract volume used during clinically indicated angiography in the cardiac catheterization laboratory.

DETAILED DESCRIPTION:
Thirty consecutive subjects who consent to participate and are undergoing planned angiography will be enrolled. The AVERT PLUS is a system which is external to the patient and connected to the control syringe that the physician uses to deliver the contrast dye to the patient. For each injection that the physician performs, the starting syringe volume, the ending syringe volume, and the net contrast delivered to the patient will be recorded. At the same time, the net volume delivered to the patient will also be recorded from the AVERT PLUS console. For each injection, these two sets of variables will be compared to determine accuracy of the AVERT PLUS to quantify net contrast volume used.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged 18 or older with cardiovascular disease scheduled to undergo clinically indicated coronary or peripheral angiography who give informed consent to participate.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with cardiovascular disease undergoing clinically indicated coronary or peripheral angiography
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Observational study of the accuracy of this system to quantify contrast volume during a clinical indicated procedure | During procedure

CONTACTS AND LOCATIONS:
Overall Officials: Michele Shepard, Study Director — Osprey Medical, Inc